CLINICAL TRIAL: NCT01331226
Title: Support Person Effectiveness Study to Promote Smoker Utilization of the QUITPLAN Helpline
Brief Title: Support Person Intervention to Promote a Smoking Helpline
Acronym: ClearWay #4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-001796; 10-008318 (Other: Mayo Clinic)
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 session telephone counseling (Experimental)
  Interventions: Behavioral: telephone counseling 3 sessions
- 1 session telephone counseling (Experimental)
  Interventions: Behavioral: telephone counseling 1 session
- written materials (Active Comparator)
  Interventions: Behavioral: written materials only

INTERVENTIONS:
Behavioral: telephone counseling 3 sessions — 3 sessions of telephone counseling
  Arms: 3 session telephone counseling
Behavioral: telephone counseling 1 session — 1 session of telephone counseling
  Arms: 1 session telephone counseling
Behavioral: written materials only — written materials only
  Arms: written materials

SUMMARY:
This study is designed to examine if a telephone-based intervention delivered to a support person (i.e., friend, spouse of a smoker) increases the smoker's use of the Minnesota helpline. In addition, the study will examine if the rate of smoker calls to the helpline is greater if the support person receives 3 intervention calls, 1 intervention call, or no calls (written materials only, control condition).

DETAILED DESCRIPTION:
We will conduct a randomized clinical trial within the ongoing service of the QUITPLAN® Helpline. Our primary aim is to examine the efficacy of two levels of telephone counseling for support persons (1 or 3 sessions) compared with a control condition on the proportion of smokers who call the Helpline over the 7 month follow-up period. We hypothesize a dose response relationship between number of telephone sessions provided to the support persons and smoker calls to the Helpline. Additional aims are to examine smoker quit attempts and cessation, and cost-effectiveness of the interventions.

Nonsmoking adult support persons (N=1020) residing in Minnesota will be enrolled and randomly assigned to one of three study conditions: (1) control condition -written self-help materials, (2) written materials plus one telephone session, or (3) written materials plus three telephone sessions. Outcome assessments will be completed by support persons and smokers at post-treatment (week 4) and at 7 month follow-up.

This design will allow for evaluation of whether results from our previous trial (Patten et al., in press, AJPM) can be replicated when the intervention is implemented within a "real-world" setting. That is all support person intervention calls will be delivered by the Helpline. Moreover, we will examine the potential efficacy and cost-effectiveness of a streamlined version of the intervention (i.e., 1 call). Furthermore, the proposed study will provide new data on quit attempts and cessation among the smokers. Ultimately, positive findings from this line of research could serve as the basis for expanding the range of helpline services to nonsmokers.

ELIGIBILITY:
Inclusion Criteria:

* The support person must

  1. reside in Minnesota
  2. be 18 years of age or older
  3. provide written informed consent
  4. be a never or former cigarette smoker (no cigarette smoking in the past 6 months)
  5. want to support a current cigarette smoker (has smoked a total of >1 cigarettes during the past 7 days) who is 18 years of age or older, resides in Minnesota, and has not been enrolled in a helpline or any other cessation program in the last 3 months
  6. be able and willing to participate in all aspects of the study
  7. have access to a working telephone
  8. have current and anticipated contact (any combination of face-to-face, telephone, text messaging, or electronic mail) with the smoker on at least 3 days a week for the 30 week study duration.

Exclusion Criteria:

* Support persons will be excluded if another support person from the same household has enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
helpline utilization | At 7 month follow-up
  smoker calls to the helpline

SECONDARY OUTCOMES:
smoker quit attempts and cessation | 7 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo CLinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Patten CA, Boyle R, Tinkelman D, Brockman TA, Lukowski A, Decker PA, D'Silva J, Lichtenstein E, Zhu SH. Linking smokers to a quitline: randomized controlled effectiveness trial of a support person intervention that targets non-smokers. Health Educ Res. 2017 Aug 1;32(4):318-331. doi: 10.1093/her/cyx050. PMID 28854569